CLINICAL TRIAL: NCT02274454
Title: Investigating the Effect of Extracellular Calcium on Oxytocin-induced Human Myometrial Contractility In-vitro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-02
Record Dates: First submitted 2014-10-09; First posted 2014-10-24 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine contraction; Oxytocin desensitization
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1.25mM Calcium-NO oxytocin pretreatment (Active Comparator)
  Interventions: Drug: Calcium
- 2.5mM Calcium-NO oxytocin pretreatment (Active Comparator)
  Interventions: Drug: Calcium
- 5.0mM Calcium-NO oxytocin pretreatment (Active Comparator)
  Interventions: Drug: Calcium
- 1.25mM Calcium-WITH oxytocin pretreatment (Active Comparator)
  Interventions: Drug: Oxytocin; Drug: Calcium
- 2.5mM Calcium-WITH oxytocin pretreatment (Active Comparator)
  Interventions: Drug: Oxytocin; Drug: Calcium
- 5.0mM Calcium-WITH oxytocin pretreatment (Active Comparator)
  Interventions: Drug: Oxytocin; Drug: Calcium

INTERVENTIONS:
Drug: Oxytocin — Experiments will be conducted with some myometrial strips pretreated with oxytocin, and others without any oxytocin pretreatment
  Other Names: pitocin
  Arms: 1.25mM Calcium-WITH oxytocin pretreatment; 2.5mM Calcium-WITH oxytocin pretreatment; 5.0mM Calcium-WITH oxytocin pretreatment
Drug: Calcium — Calcium will be applied to the myometrial strips in 3 concentrations; 1.25mM (low), 2.5mM (normal) and 5.0mM (high). Myometrial strips will be either oxytocin pretreated, or non-oxytocin pretreated.

SUMMARY:
Postpartum hemorrhage (PPH) is a leading cause of maternal morbidity and mortality worldwide and is caused most commonly by poor uterine muscle tone after delivery. The first line agent used in the prevention and treatment of PPH is oxytocin, which acts by binding with the oxytocin receptor (OTR) found on myometrial cells to cause uterine contraction. It does this by increasing levels of calcium within the myometrial cell, which promotes contraction. Women who require augmentation of labor with intravenous oxytocin because of inadequate labor progression have been shown to be at increased risk of PPH. In-vitro human myometrial models have shown that following prolonged exposure to oxytocin there is desensitization of the myometrium resulting in a significant reduction in contractility upon delivery of further oxytocin.

Optimal levels of calcium are very important for contraction of the uterine muscle. Too little calcium results in a reduced contraction. Too much calcium may result in either stronger contractions, or even possibly relaxation of the muscle and therefore a reduced contraction. The investigators currently do not know the effects of calcium on the desensitized uterine muscle.

The investigators hypothesize that myometrial contractility following desensitization of the myometrium would be reduced in myometrial samples exposed to low calcium, when compared to normal calcium or high calcium exposure. These results will help in establishing whether myometrial contraction can be augmented by increasing calcium levels within the body, or by optimizing normal physiological calcium levels, in the setting of a augmented prolonged labor, which is at higher risk of poor uterine contraction and PPH.

DETAILED DESCRIPTION:
The increased incidence of uterine atony and PPH following exogenous oxytocin administration during labor augmentation is related to myometrial OTR desensitization to oxytocin. Calcium is an important messenger required within the uterine muscle cell to result in muscle contraction following administration of oxytocin. A physiological level of calcium is known to provide optimal contractility to normal myometrium.

Characterization of the importance of low, normal or high calcium levels in a setting of prolonged exogenous oxytocin administration may provide guidance for the use of exogenous calcium as a uterotonic adjunct; or for the optimization of serum calcium levels during augmented labor. In the clinical setting of failed labor augmentation and OTR desensitization, the role of serum calcium levels is not currently known.

The investigators' previously validated in-vitro model provides a solid foundation for the study of myometrial contractility under controlled conditions, without any confounders that could be encountered in clinical settings.

The results of this study will provide insight into the effect of low, normal or high calcium levels on the oxytocin pretreated (desensitized) and non-pretreated myometrium. Based on oxytocin dose-response curves after pretreatment to oxytocin and then subsequent exposure to either low, normal or high levels of calcium, the investigators will be able to determine the role of calcium on desensitized myometrium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in this study
* Patients with gestational age 37-41 weeks
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring primary CD or first repeat CD

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who require general anesthesia
* Patients who had previous uterine surgery or more than one previous CD
* Patients with any condition predisposing to uterine atony and postpartum hemorrhage, such as abnormal placentation, multiple gestation, preeclampsia, macrosomia, polyhydramnios, uterine fibroids, bleeding diathesis, chorioamnionitis, or a previous history of postpartum bleeding
* Emergency CD in labor
* Patients on medications that could affect myometrial contractility, such as nifedipine, labetolol or magnesium sulphate.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Motility Index | 8 hours
  Motility index (MI) takes into account both the amplitude and frequency of the myometrial contraction. It is a calculated outcome, based on the formula: frequency/(10 x amplitude).
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 8 hours
  The maximum extent of uterine muscle contraction, measured in grams (g). The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 8 hours
  The number of contractions in uterine muscle (myometrium) over 10 minutes, spontaneously and in response to an agonist.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada